CLINICAL TRIAL: NCT07178600
Title: Characterization and Association of Clinical Determinants With the Occurrence of Adverse Drug Reactions Following the Administration of Tropicamide/Phenylephrine in Hospitalized Patients.
Brief Title: Clinical Determinants and Adverse Reactions to Tropicamide/Phenylephrine in Hospitalized Patients.
Acronym: RAM-TF-IOCV
Status: Recruiting | Type: Observational
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Principal Investigator, María C. Jiménez Martínez, Head of the inmunology department, Research unity, Instituto de Oftalmología Fundación Conde de Valenciana
Other Study IDs: CEI-2023/09/02; CB-042-2023 (Other: Biosafety Committee); CI-042-2023 (Other: Comité de Investigación)
Record Dates: First submitted 2025-09-11; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Adverse Drug Effect; Phenylephrine; Hypertension; Cardiovascular Complication; Ophthalmology; Ocular Discomfort
Keywords: Adverse Drug Effect; Tropicamide/phenylefrine; Tropicamide; Phenylefrine; Cardiovascular complications; Hypertension; Ophthalmology; Ocular discomfort
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Hypertension | interventions — Phenylephrine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hospitalized patients who received tropicamide/phenylephrine 8 mg/50 mg/mL.: Patients over 18 years of age who have been hospitalized to undergo a surgical procedure and who received tropicamide/phenylephrine 8 mg/50 mg/mL at the Instituto de Oftalmologia 'Conde de Valenciana' IAP
  Interventions: Drug: Ophthalmic administration of tropicamide/phenylephrine 8 mg/50 mg/mL.

INTERVENTIONS:
Drug: Ophthalmic administration of tropicamide/phenylephrine 8 mg/50 mg/mL. — Measurement of vital signs after ophthalmic administration of tropicamide/phenylephrine 8 mg/50 mg/mL

SUMMARY:
To evaluate the association between clinical determinants and the occurrence of adverse drug reactions in hospitalized patients who received tropicamide/phenylephrine 8 mg/50 mg/mL.

An ambispective, interventional, longitudinal study will be conducted to actively identify adverse reactions to tropicamide/phenylephrine 8 mg/50 mg/mL, as well as the clinical determinants that may predispose patients to the occurrence of an adverse drug reaction (ADR). Data will be collected through the administration of a questionnaire and measurement of vital signs prior to the administration of tropicamide/phenylephrine 8 mg/50 mg/mL, and subsequently at 5 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours after administration, with the aim of establishing an association between these variables.

DETAILED DESCRIPTION:
In the diagnostic approach of patients with ophthalmologic diseases, as well as for surgical purposes, the administration of mydriatic and cycloplegic drugs is indispensable. Among these, the combination of tropicamide and phenylephrine (TF) is commonly used. Studies evaluating the topical ocular administration of these medications have demonstrated an adequate risk-benefit balance; however, certain local and systemic safety aspects remain insufficiently evaluated.

Justification: This study will help identify the at-risk population (clinical determinants) prior to the administration of drugs such as TF, provide additional information regarding the safety profile of this drug at the 8 mg/50 mg/mL concentration, and propose measures to reduce the occurrence of adverse drug reactions (ADRs) in at-risk populations. It also aims to develop safety barriers that allow for safer administration of the medication. Moreover, this research provides a first approximation and establishes the basis for future studies that may compare different TF concentrations.

Hypothesis: There will be a positive association between clinical determinants and the occurrence of adverse drug reactions.

Research Question: Is there an association between the clinical determinants of hospitalized patients and the occurrence of adverse drug reactions following the administration of tropicamide/phenylephrine?

Objective: To evaluate the association between clinical determinants and the occurrence of adverse drug reactions in hospitalized patients who received tropicamide/phenylephrine 8 mg/50 mg/mL.

Materials and Methods:

An ambispective study will be conducted to identify ADRs associated with TF administration, as well as to characterize pathologies that may predispose patients to ADRs (clinical determinants, CD), through the use of a questionnaire, with the purpose of establishing an association between them.

Data Analysis:

Results will be analyzed using the Chi-square test for qualitative variables and the calculation of odds ratios (OR) with 95% confidence intervals. Quantitative variables will be analyzed using the Student's t-test for normally distributed data, or the Wilcoxon signed-rank test for data not normally distributed. Normality will be assessed with the Kolmogorov-Smirnov test (p > 0.05). The association between CDs and ADRs will be evaluated through logistic regression analysis

ELIGIBILITY:
Inclusion Criteria:

* Patients who have authorized participation in the study by signing informed consent.
* Patients over 18 years of age.
* Any sex.
* Patients from the "Instituto de Oftalmología Conde de Valenciana, IAP., sede Centro" who have been scheduled for a surgical procedure.
* Patients for whom the administration of two drops of tropicamide/phenylephrine 8 mg/50 mg/mL is indicated.
* Patients that presents any type of disease

Exclusion Criteria:

* Allergy to any component of the formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age who have been hospitalized to undergo a surgical procedure at the "Instituto de Oftalmología Conde de Valenciana, IAP".
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-09-02 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the association between clinical determinants and the occurrence of adverse drug reactions in hospitalized patients who received tropicamide/phenylephrine 8 mg/50 mg/mL. | Measurement of vital signs prior to the administration of tropicamide/phenylephrine 8 mg/50 mg/mL, and at 5 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, and 3 hours afterward.
  An ambispective, interventional, longitudinal study will be conducted to actively identify adverse reactions to tropicamide/phenylephrine 8 mg/50 mg/mL, as well as the clinical determinants that may predispose patients to the occurrence of an adverse drug reaction (ADR)
To identify and characterize the clinical determinants of hospitalized patients receiving tropicamide/phenylephrine 8 mg/50 mg/mL at the Instituto de Oftalmología Conde de Valenciana | At enrollement
  Identification of clinical determinants based on medical records review and patient interview.
To actively identify adverse reactions to tropicamide/phenylephrine 8 mg/50 mg/mL. | At enrollment Measurement of vital signs prior to the administration of tropicamide/phenylephrine 8 mg/50 mg/mL, and at 5 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, and 3 hours afterward.
  To identify adverse drug reactions (ADRs) to tropicamide/phenylephrine 8 mg/50 mg/mL through a pharmacovigilance questionnaire administered to the patient and by measuring vital signs after administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Oftalmología FAP Conde de Valenciana, IAP Sede Centro, Mexico City, Mexico Ciy, Mexico

IPD SHARING:
Plan to Share IPD: No
The plan is to share the data after finishing the protocol

REFERENCES:
- [Background] Tsui E, Sehi M, Cheng RW, Wan J, Wong T, Dorner S, Fisher JA, Hudson C. The impact of topical mydriatic ophthalmic solutions on retinal vascular reactivity and blood flow. Exp Eye Res. 2013 Jul;112:134-8. doi: 10.1016/j.exer.2013.05.005. Epub 2013 May 21. PMID 23701974